CLINICAL TRIAL: NCT00101231
Title: A Dose Escalation Study of Flavopiridol (NSC 649890) Administered as a 30 Minute Loading Dose Followed by a 4-Hour Infusion in Patients With Relapsed and Refractory Acute Leukemias
Brief Title: Flavopiridol in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia, Acute Lymphoblastic Leukemia, or Chronic Myelogenous Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01461; OSU 0479; NCI-6947; OSU-2004C0085; OSU-0479; CDR0000404374; U01CA076576 (NIH)
Record Dates: First submitted 2005-01-07; First posted 2005-01-10 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Adult Acute Basophilic Leukemia; Adult Acute Eosinophilic Leukemia; Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Blastic Phase Chronic Myelogenous Leukemia; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Relapsing Chronic Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Basophilic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute; Blast Crisis; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — alvocidib

ARMS (1):
- Treatment (flavopiridol) (Experimental): Patients receive flavopiridol IV over 30 minutes followed by a 4-hour infusion on days 1-3. Treatment repeats every 21 days for up to 6 courses in the absence of unacceptable toxicity or disease progression.
  Interventions: Drug: alvocidib

INTERVENTIONS:
Drug: alvocidib — Given IV
  Other Names: FLAVO; flavopiridol; HMR 1275; L-868275

SUMMARY:
This phase I trial is studying the side effects and best dose of flavopiridol in treating patients with relapsed or refractory acute myeloid leukemia, acute lymphoblastic leukemia, or chronic myelogenous leukemia. Drugs used in chemotherapy, such as flavopiridol, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximal tolerable dose of flavopiridol in relapsed or refractory acute leukemia in adults (Stratum 1) and children (Stratum 2).

II. To define the qualitative and quantitative toxicities of flavopiridol in regard to organ specificity, time course, predictability, and reversibility.

III. To determine the preliminary clinical activity of flavopiridol in adults (Stratum 1) and children (Stratum 2) using this novel schedule in acute leukemia.

IV. To evaluate the plasma and cellular pharmacokinetics of flavopiridol in patients enrolled on this study.

SECONDARY OBJECTIVES:

I. To measure pharmacodynamic measurements including effects on cell cycle; down modulation of bcl-2, mcl-1, XIAP, bax, RNA polymerase II phosphorylation; and signaling via the VEGF (VEGF, VEGF-R1, VEGF-R2, HIF-1), NF-Kappa B pathway, and PI3kinase pathway; and correlate with Css and other pharmacokinetic features.

II. To assess drug induced apoptosis of acute leukemia cells in vitro and subsequent relationship to clinical response based upon Css of flavopiridol attained in vivo.

II. To determine if increase in inflammatory cytokines (TNF-alpha, gamma-IFN, IL-6 and IL-8) correlate with pharmacokinetics, pharmacodynamics, laboratory (decrease in serum albumin) and clinical (hypotension observed with the first administration of flavopiridol) parameters of treatment.

OUTLINE: This is a dose-escalation study. Patients are stratified according to age group (adult [≥ 18 years] vs pediatric [1-17 years]).

Patients receive flavopiridol intravenously (IV) over 30 minutes followed by a 4-hour infusion on days 1-3. Treatment repeats every 21 days for up to 6 courses in the absence of unacceptable toxicity or disease progression. Cohorts of 3-6 patients receive escalating doses of flavopiridol until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed up every 2 months for 1 year and then every 6 months for 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of one of the following:

  * Acute myeloid leukemia (AML) or acute lymphoblastic leukemia (ALL) meeting 1 of the following criteria:

    * Refractory to initial treatment (stratum 1)
    * Recurrent disease after prior high-dose chemotherapy with or without stem cell support (stratum 1)
    * High-risk refractory disease defined as failed ≥ 2 regimens for remission induction (i.e., twice induction failure) (stratum 2)
    * High-risk relaspsed disease defined as disease in second or greater bone marrow relapse (stratum 2)
  * Chronic myelogenous leukemia in blast crisis (stratum 1)

    * Myeloid or lymphoid blast crisis that did not respond to or progressed after prior high-dose imatinib mesylate (600-800 mg/day for ≥ 2 weeks)
* No acute promyelocytic leukemia
* Ineligible for or unwilling to undergo potentially curative allogeneic or autologous stem cell transplantation

  * Patients with relapsed AML that is refractory to re-induction therapy comprising an active, intensive salvage regimen are eligible
* CNS involvement allowed provided there are no residual leukemic cells in the cerebrospinal fluid after intrathecal chemotherapy or radiotherapy
* Performance status - ECOG ≥ 2 for patients > 10 years of age
* Performance status - Lansky 50-100% for patients ≤ 10 years of age
* At least 8 weeks
* Bilirubin ≤ 2 times upper limit of normal (ULN)* (unless due to Gilbert's syndrome)
* ALT and AST ≤ 5 times ULN*
* Creatinine ≤ 2.0 mg/dL* (stratum 1)
* Creatinine > 1.3 times ULN (stratum 2)
* LVEF ≥ 40% by echocardiogram or MUGA (stratum 1)
* Shortening fraction ≥ 28% by echocardiogram (stratum 2)
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No history of allergy to study drug
* No active infection requiring IV antibiotics
* No serious medical or psychiatric illness that would preclude giving informed consent or limit survival
* No other uncontrolled illness
* See Disease Characteristics
* Recovered from all prior immunotherapy treatment-related toxicity (stratum 2)
* More than 8 weeks since prior biological agents (e.g., monoclonal antibodies) (stratum 2)
* See Disease Characteristics
* Recovered from all prior chemotherapy treatment-related toxicity (stratum 2)
* More than 24 hours since prior hydroxyurea (for patients who do not have highly proliferative disease)*
* More than 2 weeks since other prior chemotherapy (6 weeks for nitrosourea or mitomycin)
* No other concurrent chemotherapy
* Prior hydrea and/or steroids allowed (stratum 2)
* No concurrent hormones, except steroids for adrenal failure or infusional toxicity (i.e., cytokine release syndrome) or hormones for non-disease-related conditions (e.g., insulin for diabetes)
* See Disease Characteristics
* Recovered from all prior radiotherapy treatment-related toxicity (stratum 2)
* More than 2 weeks since prior radiotherapy
* No concurrent palliative radiotherapy
* Post stem cell transplant allowed provided completion ≥ 4 months prior to study entry and no evidence of active acute or chronic graft vs host disease (stratum 2)
* No other concurrent investigational agents
* No concurrent chronic systemic anticoagulant therapy for a medical condition (e.g., deep vein thrombosis or atrial fibrillation)

  * Concurrent heparin allowed to maintain central line patency (i.e., catheter flush)
* No other concurrent anticancer therapy

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2004-10; Primary Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Maximal tolerable dose of flavopiridol | Day 21

CONTACTS AND LOCATIONS:
Overall Officials: William Blum, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Derived] Blum W, Phelps MA, Klisovic RB, Rozewski DM, Ni W, Albanese KA, Rovin B, Kefauver C, Devine SM, Lucas DM, Johnson A, Schaaf LJ, Byrd JC, Marcucci G, Grever MR. Phase I clinical and pharmacokinetic study of a novel schedule of flavopiridol in relapsed or refractory acute leukemias. Haematologica. 2010 Jul;95(7):1098-105. doi: 10.3324/haematol.2009.017103. Epub 2010 May 11. PMID 20460644